CLINICAL TRIAL: NCT06832384
Title: Intensive Physiotherapy Intervention in Children Affected by Tumors Located in Posterior Cranial Fossa
Brief Title: Intensive Physiotherapy in Children Affected by Posterior Fossa Tumors
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 21.2022 Oss
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Posterior Fossa Tumor
MeSH Terms: conditions — Infratentorial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group
  Interventions: Procedure: intensive physiotherapy

INTERVENTIONS:
Procedure: intensive physiotherapy — the dosing of the intensive physiotherapy is of 2 sessions a day, lasting 45 minutes each, administered 5 days a week, for a period of 4 weeks.
  the physiotherapy is mainly addressed to the improvement of gross motor movement and balance and the training is designed according to the specific need of the subject recruited. it is not allowed the use of technological devices, excepted treadmill training.

SUMMARY:
The objective of the current study is to describe the effectiveness of conventional and intensive physiotherapeutic intervention in improving gross motor skills (i.e. postural changes, walking and balance skills) in children affected by posterior fossa tumors

DETAILED DESCRIPTION:
The surgery aimed to remove tumors located in the cranial posterior fossa can lead, as a consequence, to a clinical condition of ataxia.

Children affected by this condition are commonly referred to physiotherapy treatment, even though the level of scientific evidence in the field of motor rehabilitation is still lacking.

The objective of the current study is to describe the effectiveness of conventional and intensive physiotherapeutic intervention in improving gross motor skills (i.e. postural changes, walking and balance skills) in children affected by posterior fossa tumors.

By conventional physiotherapy intervention we mean a therapeutic path with a 1:1 operator-patient ratio and which does not make use of robotic or virtual reality devices.

By intensive we mean that it occurs twice a day, 5 days a week, for a duration of four weeks.

Given the high variability in the severity of the clinical pictures, the primary objective will be the patient's improvement in gross motor skills as a whole, which will be identified with the Gross Motor Function Measurment (GMFM) scale.

Changes will also be monitored with respect to the autonomy and assistive care in the daily life of the recruited patients (scored through WeeFIM or FIM), the risk of fall (scored through the Pediatric Balance Scale) and with a sign-specific scale on ataxia (Scale for Assessment and Rating of Ataxia) Finally, for walking patients, walking resistance will be assessed through the 6 minute walking test (6MWT)

ELIGIBILITY:
Inclusion Criteria:

* subjects who underwent to surgical resection of tumors located in posterior fossa, age between 0 and 25 years

Exclusion Criteria:

* Subjects that are currently addressed to rehabilitative protocols availing of technological devices

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, teen agers and young adults affected by posterior fossa tumors will be collected in three different centers, nemely IRCCS Medea located in Bosisio Parini, Conegliano and Brindisi.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) | A first assessment is provided at the enrollment and the second assessment is administered at the end of the treatment, after 4 weeks
  The GMFM is composed by 88 items (providing a range of score form 0 to 3 each) divided in 5 sections: A- lying and rolling; B- sitting; (C) crawling and kneeling; D - standing; E - walking, running and jumping.
  The total score can range between 0 (subject can't perform any gross motor activity) to a maximum of 264 (the subject completely developed his gross motor skills).

SECONDARY OUTCOMES:
Six minutes walking test (6MWT) | A first assessment is provided at the enrollment and the second assessment is administered at the end of the treatment, after 4 weeks
  The test is used to evaluate the walking endurance. During the test the distance covered over six minute of self-paced walking along a standardized path is measured, providing a reliable measure of patient's limitations as community ambulators.
Scale for the Assessment and Rating of Ataxia (SARA) | A first assessment is provided at the enrollment and the second assessment is administered at the end of the treatment, after 4 weeks
  This scale is developed to quantify the severity of the ataxia. It includes motor tasks (that investigate the most common deficits, like imbalance, tremors, dysmetria, rhythmic movements) and one item that examine the speech. This validated tool scores from 0 (no ataxia) to 40 (severe ataxia) and is composed by 8 items that comprise assessment of speech, upper and lower limb ability
Pediatric Balance Scale (PBS) | A first assessment is provided at the enrollment and the second assessment is administered at the end of the treatment, after 4 weeks
  The scale is used to assess balance skills in school-aged children. The scale consists of 14 balance-related test items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
WeeFIM | A first assessment is provided at the enrollment and the second assessment is administered at the end of the treatment, after 4 weeks
  This assessment measures the type and amount of assistance required for a person with a disability to perform basic life activities effectively.
  It is an 18-item performance measurement system that documents self-care, functional mobility, and cognitive abilities. The self-care domain includes 8 items (eating, grooming, bathing, lower and upper body dressing, toileting, as well as bowel and bladder control). The mobility domain includes 5 items (chair, toilet, and tub transfers, walking or wheelchair management, and stairs). The cognitive domain includes 5 items (language comprehension and expression, social interaction, problem solving, and memory).
gait analysis | A first assessment is provided at the enrollment and the second assessment is administered at the end of the treatment, after 4 weeks
  3D gait analysis is an assessment performed with an eight cameras optoelectronic system working at 100 Hz and two force plates. During the analysis participants are asked to walk at their preferred speed and barefoot. For each assessment, at least five trials for the left and the right limbs were collected and processed using dedicated software. The most representative trial for each child is selected for further analysis.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS E. Medea, Brindisi, Brindisi
  - IRCCS E. Medea, Bosisio Parini, Lecco
  - IRCCS E. Medea, Conegliano, Treviso

IPD SHARING:
Plan to Share IPD: Undecided